CLINICAL TRIAL: NCT06180421
Title: Development of the Mitochondrial Video Assessment (MVA) as an Outcome Measure for the Evaluation of Patients With Mitochondrial Myopathies
Brief Title: Mitochondrial Video Assessment Source Material Study
Status: Completed | Type: Observational
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: United Mitochondrial Disease Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAS-CAS009
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: PolG, Primary Mitochondrial Myopathy
Keywords: PoIG; Primary Mitochondrial Myopathy; MELAS; CPEO
MeSH Terms: conditions — MELAS Syndrome; Ophthalmoplegia, Chronic Progressive External

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PolG: Genetically confirmed PoLG patients 16 years or older
- PMM: Genetically confirmed Primary Mitochondrial Myopathy patients 16 years or older

SUMMARY:
Source material collection of videos to develop the Mitochondrial Video Assessment (MVA) for patients with mitochondrial myopathies.

DETAILED DESCRIPTION:
This observational research is being conducted to facilitate the development of 2 related, disease-specific outcome measures assessing ease of movement in PMM and PolG clinical trials. The Mitochondrial Video Assessment (MVA) utilizes remote video capture to assess subtle shifts in compensatory movement patterns and measure change in function over time, and the Current State Questionnaire asks participants about external factors in their daily lives which may influence fluctuations in their symptoms. As part of the questionnaire, participants are asked to rate their own perception of their functional ability using a Patient Global Impression of Severity (PGI-S) scale.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old and above
* Confirmed diagnosis of PMM or PolG
* Ability to understand and speak English
* Ability and willing to consent
* Able and willing to participate and perform tasks while being recorded
* Designating a recording partner to assist with video captures is strongly advised, but not required

Exclusion Criteria:

* N/A

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons aged 16 and older living with a confirmed diagnosis of PMM or PoIG.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Source Material Videos | 2 weeks
  Initiate feasibility testing and collect source material videos from patients with Primary Mitochondrial Myopathy (PMM, n=35) or a PolGamma (PolG) mutation (n=15) to facilitate development of the Mitochondrial Video Assessment (MVA).

SECONDARY OUTCOMES:
PGI-S | 2 weeks
  Identify external factors which may influence participant performance on functional assessments and collect Patient Global Impression of Severity (PGI-S) at the time of each capture to facilitate the development of a patient-reported Current State Questionnaire to be deployed in conjunction with the MVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Casimir, Kingston, Massachusetts, United States

REFERENCES:
- [Background] Rajakulendran S, Pitceathly RD, Taanman JW, Costello H, Sweeney MG, Woodward CE, Jaunmuktane Z, Holton JL, Jacques TS, Harding BN, Fratter C, Hanna MG, Rahman S. A Clinical, Neuropathological and Genetic Study of Homozygous A467T POLG-Related Mitochondrial Disease. PLoS One. 2016 Jan 6;11(1):e0145500. doi: 10.1371/journal.pone.0145500. eCollection 2016. PMID 26735972
- [Background] Stumpf JD, Saneto RP, Copeland WC. Clinical and molecular features of POLG-related mitochondrial disease. Cold Spring Harb Perspect Biol. 2013 Apr 1;5(4):a011395. doi: 10.1101/cshperspect.a011395. PMID 23545419
- [Background] Gorman GS, Schaefer AM, Ng Y, Gomez N, Blakely EL, Alston CL, Feeney C, Horvath R, Yu-Wai-Man P, Chinnery PF, Taylor RW, Turnbull DM, McFarland R. Prevalence of nuclear and mitochondrial DNA mutations related to adult mitochondrial disease. Ann Neurol. 2015 May;77(5):753-9. doi: 10.1002/ana.24362. Epub 2015 Mar 28. PMID 25652200
- [Background] Goldstein A, Rahman S. Seeking impact: Global perspectives on outcome measure selection for translational and clinical research for primary mitochondrial disorders. J Inherit Metab Dis. 2021 Mar;44(2):343-357. doi: 10.1002/jimd.12320. Epub 2020 Oct 29. PMID 33016339
- [Background] Pitceathly RDS, Keshavan N, Rahman J, Rahman S. Moving towards clinical trials for mitochondrial diseases. J Inherit Metab Dis. 2021 Jan;44(1):22-41. doi: 10.1002/jimd.12281. Epub 2020 Sep 2. PMID 32618366
- [Background] Rahman S, Copeland WC. POLG-related disorders and their neurological manifestations. Nat Rev Neurol. 2019 Jan;15(1):40-52. doi: 10.1038/s41582-018-0101-0. PMID 30451971
- [Background] Instrustry FGf. Patient-Focused Drug Development: Methods to Identify What is Important to Patients. 2022.
- [Background] Industry FGf. Methods to Identify What is Important to Patients and Select, Develop, and Modify Fit-for-Purpose Clinical outcomes Assessments. 2018.